CLINICAL TRIAL: NCT02762968
Title: The Effects of 8-weeks of Probiotic and HMB Supplementation on Immune and Digestive Function in Special Operations Soldiers
Brief Title: The Effects of Probiotic and HMB Supplementation on Immune and Digestive Function in Special Operations Soldiers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metabolic Technologies Inc. (Industry)
Collaborators: University of Central Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MTI2016-CS02
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Military Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo capsules similar to the experimental treatments.
  Interventions: Dietary Supplement: Placebo
- HMB (Experimental): HMB capsules providing 3 g of calcium HMB per day.
  Interventions: Dietary Supplement: HMB
- HMB + BC30 (Experimental): Capsules providing 3 g calcium HMB per day plus Bacillus Coagulans GBI-30, 6086 (BC30) mixed in water.
  Interventions: Dietary Supplement: HMB; Dietary Supplement: BC30

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo capsules similar to the experimental treatments.
  Arms: Placebo
Dietary Supplement: HMB — Capsules containing calcium HMB.
  Arms: HMB; HMB + BC30
Dietary Supplement: BC30 — Bacillus Coagulans GBI-30, 6086 (BC30) mixed in water.
  Arms: HMB + BC30

SUMMARY:
The study will determine whether acute ingestion of a probiotic combined with beta-hydroxy-beta-methylbutyrate (HMB) can enhance immune and digestive function in soldiers during 8-weeks of advanced infantry training.

DETAILED DESCRIPTION:
Up to sixty soldiers from an elite infantry unit will perform a parallel design investigation. Soldiers will be randomly assigned to one of four groups. Group 1 will consume the probiotic plus HMB, group 2 will consume HMB only, group 3 will consume only the probiotic, and group 4 will consume only placebo. All four groups will be garrisoned together, eat the same meals, and perform the same activity. All groups will be tested before as well as after an 8-week advanced infantry training program. During each testing session resting blood samples will be obtained to assess cytokine, inflammatory, and muscle damage markers. Additionally, questionnaires will be used to determine digestive health. Anthropometric, performance, and muscle volume measures will also be assessed prior to and immediately following the supplementation and training protocol.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Member of the same unit of the IDF

Exclusion Criteria:

* Current use of dietary supplements
* Current chronic use of medications

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2016-04; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Maintenance of Immune function | 8 weeks
  Immune function assessed by blood biochemical analysis (ELISA).

SECONDARY OUTCOMES:
Maintenance of Digestive Function | 8 Weeks
  Digestive function assessed by questionnaire.
Maintenance of Muscle Volume | 8 Weeks
  Muscle volume will be assessed using a 3.0 Tesla whole-body imager (cubic centimeter)

CONTACTS AND LOCATIONS:
Overall Officials: Jay R Hoffman, PhD, Study Director — University of Cenral Florida
Locations (1):
- Israel, Beersheva, Israel

IPD SHARING:
Plan to Share IPD: No